CLINICAL TRIAL: NCT05680181
Title: Multicenter National Observational and Prospective Study of a Cohort of Children With Molluscum Contagiosum (MC) Treated With a 5% Solution of Potassium Hydroxide (Molutrex®) Applied Locally to the Skin
Brief Title: Study of a Cohort of Children With Molluscum Contagiosum (MC) Treated With a 5% Solution of Potassium Hydroxide (Molutrex®) Applied Locally to the Skin
Acronym: SERENITE
Status: Completed | Type: Observational
Sponsor: Laboratoire Dermatologique ACM (Industry)
Collaborators: Clin-Experts (Industry)
Responsible Party: Sponsor
Other Study IDs: 2022-A01503-40
Record Dates: First submitted 2022-12-16; First posted 2023-01-11 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Molluscum Contagiosum
Keywords: Molluscum Contagiosum; Observational study; Medical device
MeSH Terms: conditions — Molluscum Contagiosum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Molutrex® a 5% potassium hydroxide solution for topical application to the skin. Molutrex® is intended for the superficial treatment of certain types of warts, molluscum contagiosum and is composed of potassium hydroxide (5%) purified water. With regard to the 2017/745 RDM, he is a class IIa medical device. In accordance with Regulation (EU) 2017/745 of the European Parliament and of the Council of April 5, 2017 relating to medical devices, as part of the Molutrex® Post-Marketing Monitoring Plan, the objective of this study is to have data on the performance , safety and suitability for real-life use of Molutrex® in a prospective cohort of patients with molluscum contagiosum.

Since molluscum contagiosum is most prevalent in children, and potassium hydroxide is used very little in adults (because most often they are immunocompromised patients requiring other antiviral treatments), the study will be conducted in children aged 2 to 10 years. This population represents the majority of patients treated with Molutrex®, although the product can be used in adults. The study includes 2 visits, the objective of the study being to evaluate the percentage of children healed at 45 days, healing defined by a reduction of more than 90% in the number of lesions present at inclusion in the study.

ELIGIBILITY:
Inclusion Criteria:

Child aged 2 to 10 years old :

* Ambulatory
* Seen in dermatology consultation for molluscum contagiosum
* For which a treatment with a 5% solution of potassium hydroxide (Molutrex®) in local cutaneous application has been decided by the dermatologist as monotherapy
* Not treated for their molluscum contagiosum in the previous month
* For which one of the parents gives their written consent to participate

Exclusion Criteria:

Doubt about the diagnosis of molluscum contagiosum Molluscum contagiosum surge already treated Immunocompromised child Atopic eczema in outbreak Lesions around the eye

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Child seen in private dermatology consultation for suspected molluscum contagiosum
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2023-01-20 (Actual); Primary Completion 2024-01-26 (Actual); Study Completion 2024-01-26 (Actual)

PRIMARY OUTCOMES:
Percentage of children healed healing defined by a decrease of more than 90% in the number of lesions present at D0. | at day 45 +- 2 days

SECONDARY OUTCOMES:
Percentage change in the number of lesions compared to D0 | at day 45 +- 2 days
Percentage of patients according to the reduction in the number of lesions compared to D0 | at day 45 +- 2 days
  (> 90%, 90% 75%; 74%-50%; 49%-25%; < 25%)
Percentage of children in whom new lesions appeared since inclusion according to the parents | at day 45 +- 2 days
Time of disappearance of the initial lesions (judgment of the parents) | up to 45 days
Disappearance of pruritus since inclusion | at day 45 +- 2 days
  Yes/non Yes/no
Occurrence of contamination of a subject of the family since inclusion | at day 45 +- 2 days
  Yes/no
Compliance with the terms of use of the prescribed treatment | at day 45 +- 2 days
  Yes/no
Assessment of the ability to use the treatment | at day 45 +- 2 days
  Assessed with 4 questions :
  Did you find the instructions easy or difficult to understand (Very difficult;Difficult;Neither easy nor difficult;Easy;Very easy) Did you find the bottle easy or difficult to open (Very difficult;Difficult;Neither easy nor difficult;Easy;Very easy) Did you find the product easy or difficult to apply (Very difficult;Difficult;Neither easy nor difficult;Easy;Very easy) Did you find the bottle with the cap with the brush easy or difficult to close (Very difficult;Difficult;Neither easy nor difficult;Easy;Very easy)
Assessment of tolerance | at day 45 +- 2 days
  Tolerance is measured by adverse events reported

CONTACTS AND LOCATIONS:
Overall Officials: Eric CAUMES, Principal Investigator — Hôtel Dieu de Paris
Locations (1):
- Multiple locations, Multiple Locations, France

IPD SHARING:
Plan to Share IPD: Undecided